CLINICAL TRIAL: NCT04442035
Title: Clinical Efficacy Study on 5-element Music Therapy on Patients With Physically and Psychologically Unbalance After Breast Cancer Surgery
Brief Title: 5-element Music Therapy on Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2016-043-01
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer Female; Quality of Life; Depression, Anxiety
Keywords: breast cancer; music therapy; Quality of Life; Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The teatment group (Experimental): 5-element misic therapy
  Interventions: Behavioral: 5-element music therapy
- The control group (Experimental): health education
  Interventions: Behavioral: 5-element music therapy

INTERVENTIONS:
Behavioral: 5-element music therapy — participants were treated by TCM five-phase music therapy for not less than 30 minutes per day, and group music therapy was performed every three weeks. In addition, the therapeutic schedule is composed of treatment time (1pm-2pm, 9pm-11pm), frequency treatment (two times a day), intervention (10-15 minutes in the afternoon, 30 minutes in the evening) and content (individuals: dialectical selection of music; groups: community singing, every three weeks).
  Other Names: health education

SUMMARY:
In this study, we observed the clinical effect of using music therapy of TCM to improve the status of liver depression in patients with postoperative breast cancer patients, Second we want to explore the efficacy and advantages of traditional Chinese medicine in patients with postoperative breast cancer, and to reveal the clinical use of the efficacy and superiority.

DETAILED DESCRIPTION:
The study is a prospective controlled trial. Sixty-four patients were divided randomly into two groups. Patients were randomly divided into the treatment group and the control group, namely, the music treatment group and the health education group. The treatment group was given at least 30 minutes of individual music therapy and group music therapy every 3 weeks. Instead, the control group was given every 3 weeks of health education preach. It will take 12 weeks for treatment and observation. The efficacy was evaluated by observing the beginning and end of the trial of the Self-Rating Anxiety Scale score, the Self-Rating Depression Scale score, and the Breast Cancer Patients' Quality of Life Scale. At the end of the treatment, we take software packages SPSS 20.0 for management and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of breast cancer in clinical stage (Ⅰ, Ⅱ, Ⅲ) and postoperative breast cancer during one month;
* All participants had to have clinical depression and stagnation of liver qi;
* age 27-66;
* participants are conscious and willing to be followed up during the treatment.

Exclusion Criteria:

* Metastasis of breast cancer or serious complications;
* Patients with major depressive disorder;
* The past medical history of mental disorders;
* The primary diseases including liver, kidney, cerebrovascular, cardiovascular and hematopoietic system diseases;
* Participating in another clinical study or undergoing another intervention;
* Patients with hearing loss.

Ages: 27 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-06-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Self-Rating Anxiety Scale (SAS) score at 3 Months | Baseline and months 3
  The SAS is validated,self-reported table assessing anxiety state over the past 3 month.Possible scores below 50 defined as no anxiety,range 50 to 59 is Mild anxiety,range 60 to 69 is Moderate anxiety , scores above 70 is Severe Anxiety.The higher the score the worse state change=( months 3 score -Baseline score )
Change From Baseline in Self-Rating Depression Scale(SDS) score at 3 Months | Baseline and months 3
  The SDS is validated,self-reported table assessing depression state over the past 3 month.Possible scores below 52 defined as no anxiety,range 53 to 62 is Mild anxiety,range 63 to 72 is Moderate anxiety , scores above 73 is Severe Anxiety.The higher the score the worse state change=( months 3 score -Baseline score )
Change From Baseline in Quality of Life (FACT-B score) at 3 Months | Baseline and months 3
  The FACT-B is validated,self-reported table assessing quality of life over the past 3 month. The scale evaluation breast cancer patient's quality of life for 5 - dimensional such as physiological, social&family, emotions ; status ; breast cancer additional entries .
  The higher the score , the better state change=( months 3 score -Baseline score )

CONTACTS AND LOCATIONS:
Overall Officials: Zheng zhuanfang, Study Chair — Second Clinical College of Guangzhou University of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Chinese medicine hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No